CLINICAL TRIAL: NCT01766895
Title: Long-term Follow Up of Viral Hepatitis in Uremic Patients in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUH-IRB-980083; 100CM-KMU-09 (Other Grant/Funding Number: KMUH)
Record Dates: First submitted 2013-01-01; First posted 2013-01-11 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Uremia; Viral Hepatitis
Keywords: uremia; HBV; HCV; seroclearance
MeSH Terms: conditions — Uremia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — host factors ssociated with viral hepatitis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- uremic patients: blood sampling of viral hepatitis in uremic patients
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — blood sampling of viral hepatitis to determined seroprevalence in uremic patients

SUMMARY:
The linkage between viral hepatitis and renal failure is complex. The current study aims to exlore the long-term prevalence of viral hepatitis among uremic patients in Taiwan

DETAILED DESCRIPTION:
Patients are prospectively recruited from 15 hemodialysis units including one medical center, 3 satellite hospitals and 11 local clinics in Taiwan. Patients who provided informed consents for blood tests including genetic study related to HCV spontaneous seroclearance are enrolled for analysis. All the eligible subjects are tested for both HCV antibodies (third-generation, enzyme immunoassay; Abbott Laboratories, North Chicago, IL) and hepatitis B surface antigen (HBsAg). HCV RNA is tested by polymerase chain reaction (Cobas Amplicor Hepatitis C Virus Test, V.2.0; Roche Diagnostics, Branchburg, New Jersey, USA; detection limit: 50 IU/ml) twice for at least 6 months apart if anti-HCV is positive to ensure chronicity of HCV infection. HBsAg is quantified with the use of a standard quantitative chemiluminescent microparticle immunoassay (ARCHITECT HBsAg, Abbott Diagnostics). The concentration of HBsAg in the specimen is determined using a previously generated Architect HBsAg calibration curve (range, 0.05-250 IU/mL). Samples with serum HBsAg titer >250 IU/mL were diluted at 1:20 and 1:500 with the Architect HBsAg diluent and retested to expand the upper limit of the dynamic range from 250 to 125,000 IU/mL. Serum HBV DNA is determined by a standardized automated quantitative PCR assay (Cobas Amplicor HBV Monitor; Roche Diagnostics; detection limit 200 copies/ml) if patients are seropositive for HBsAg.

ELIGIBILITY:
Inclusion Criteria:

* uremic patients

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Uremic patients will recruited from 15 hemodialysis units including one medical center, 3 satellite hospitals and 11 local clinics in Taiwan.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
seroprevalence of viral hepatitis in uremic patients | 10 years

SECONDARY OUTCOMES:
factors associated with HCV clearance or reappearance | 10 years

OTHER OUTCOMES:
HBV seroconversion | 10 years
  Factors assocaited with HBV seroconversion

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Feng Huang, M.D., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Wei YJ, Hsu PY, Lee JJ, Niu SW, Huang JC, Hsu CT, Jang TY, Yeh ML, Huang CI, Liang PC, Lin YH, Hsieh MY, Hsieh MH, Chen SC, Dai CY, Lin ZY, Chen SC, Huang JF, Chang JM, Hwang SJ, Chuang WL, Huang CF, Chiu YW, Yu ML. Evolutionary seroepidemiology of viral hepatitis and the gap in hepatitis C care cascades among uraemic patients receiving haemodialysis in Taiwan-the Formosa-Like Group. J Viral Hepat. 2021 May;28(5):719-727. doi: 10.1111/jvh.13477. Epub 2021 Feb 13. PMID 33533547